CLINICAL TRIAL: NCT02263898
Title: Biomarkers of Durable Response With Intermittent Therapy With LGX818 and MEK162 Combined Therapy in Patients With BRAF Mutant Metastatic Melanoma
Brief Title: Intermittent LGX818 and MEK162 in Treating Patients With Metastatic Melanoma Who Have BRAFV600 Mutations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: closed without enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-000616; NCI-2014-01971 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-000616 (Other: Jonsson Comprehensive Cancer Center); P01CA168585 (NIH)
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2016-12

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (LGX818, MEK162) (Experimental): Patients receive LGX818 PO QD and MEK162 PO BID continuously for 8 weeks followed by intermittent dosing in subsequent cycles (3 weeks off therapy, 5 weeks on therapy). Cycles repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Raf kinase inhibitor LGX818; Drug: binimetinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Raf kinase inhibitor LGX818 — Given PO
  Other Names: LGX818
Drug: binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK inhibitor ARRY-438162; MEK162
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies intermittent dosing of BRAF inhibitor LGX818 (encorafenib) and MEK inhibitor MEK 162 (binimetinib) in treating patients with melanoma that has spread to other parts of the body (metastatic) and have a BRAF V600 mutation. LGX818 and MEK162 may stop the growth of tumor cells by blocking different enzymes needed for cell growth. Giving LGX818 and MEK162 with breaks between each course (intermittently) may help delay the time when tumors become resistant to the drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. One year progression free survival (PFS) rate.

SECONDARY OBJECTIVES:

I. Obtain biopsy samples from patients treated with an intermittent schedule of LGX818 and MEK162 to study adaptive and acquired resistance as well as melanoma evolutionary patterns.

II. Study molecular changes of adaptive resistance and acquired resistance to LGX818 and MEK162 in circulating melanoma cells.

III. Study plasma samples for circulating deoxyribonucleic acid (DNA), microribonucleic acid (microRNA) and protein signatures of adaptive resistance and acquired resistance.

IV. Explore the median progression free survival and overall survival of patients receiving an intermittent schedule of LGX818 and MEK162.

OUTLINE:

Patients receive LGX818 orally (PO) once daily (QD) and MEK162 PO twice daily (BID) continuously for 8 weeks, followed by intermittent dosing in subsequent cycles (3 weeks off therapy, 5 weeks on therapy). Cycles repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically confirmed diagnosis of metastatic melanoma with the presence of the B-Raf proto-oncogene, serine/threonine kinase (BRAFV600) mutation
* Eastern Cooperative Oncology Group (ECOG) performance status < 3
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dL without transfusions
* Platelets (PLT) >= 90 x 10^9/L without transfusions
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN); patient with liver metastases =< 5 x ULN
* Total bilirubin =< 2 x ULN, or < 5 ULN if Gilbertâ€™s disease
* Creatinine =< 1.5 mg/dL, or calculated creatinine clearance (determined as per Cockcroft-Gault) >= 50 mL/min
* Left ventricular ejection fraction (LVEF) >= 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram (ECHO)
* Corrected QT (QTc) interval =< 480 ms
* Able to take oral medications
* Patient is deemed by the Investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up)
* Negative serum beta (Î²) human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within 72 hours prior to first dose

Exclusion Criteria:

* Prior exposure to BRAF or MEK inhibitors
* Any active central nervous system (CNS) lesion (i.e., those with radiographically unstable, symptomatic lesions) and/or leptomeningeal metastases; however, patient treated with stereotactic radiotherapy, whole brain radiation or surgery are eligible if patient remained without evidence of CNS disease progression >= 4 weeks; patients must be off corticosteroid therapy for >= 2 weeks
* History or current evidence of retinal vein occlusion (RVO) or predisposing factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* History of retinal degenerative disease
* History of Gilbertâ€™s syndrome
* Previous or concurrent malignancy is not an exclusion provided that the other malignancy is considered under control and target lesions from melanoma are clearly defined for response assessment
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) < 6 months prior to screening,
  * Symptomatic chronic heart failure, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia
* Uncontrolled arterial hypertension despite medical treatment
* Known positive serology for HIV (human immunodeficiency virus), active hepatitis B, and/or active hepatitis C infection
* Patients who have neuromuscular disorders that are associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment; muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on MEK162 treatment
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Patients taking non-topical medication known to be a strong inhibitor of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); however patients who either discontinue their treatment or switch to another medication at least three days prior to randomization are eligible
* Any other condition that would, in the Investigatorâ€™s judgment, contraindicate the patientâ€™s participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/psychological issues, etc.
* Patients who have undergone major surgery =< 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation; highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening); for female patients on the study, the vasectomized male partner should be the sole partner for that patient
  * Combination of any of the two following (a+b or a+c or b+c)

    * a. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
    * b. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * c. Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * In case of use of oral contraception, women should have been stable on the same pill before taking study treatment
  * Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception
  * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse while taking the drug and for 8 weeks after stopping treatment and should not father a child in this period; a condom is required to be used also by vasectomized men
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PFS rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States